CLINICAL TRIAL: NCT00104143
Title: A Randomized, Double-blind, Placebo Controlled Dose-ranging Study to Determine the Effect on MRI Lesions and Safety of A4I Antagonist in Relapsing Multiple Sclerosis.
Brief Title: A Study of A4I Antagonist in Patients With Relapsing Multiple Sclerosis.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN18344
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Drug: A4I Antagonist

SUMMARY:
This study will compare the effect of A4I antagonist and placebo on MRI lesions,on clinical endpoints, and safety in patients with relapsing Multiple Sclerosis (MS). Eligible patients will be randomized to receive placebo or A4I antagonist, 20mg, 80mg or 300mg, po bid. Patients will undergo MRI brain scans and MS clinical evaluations at intervals throughout the study. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-59 years of age;
* relapsing multiple sclerosis patients with types 1-4 (established through McDonald criteria);
* >=1 MS attack or a Gd-enhancing MRI lesion between 1 month and 1 year before enrollment;
* EDSS score of <=6.5;
* inadequate response to approved treatment(Canada only).

Exclusion Criteria:

* MS attack within 1 month before enrollment;
* systemic corticosteroids within 1 month before enrollment;
* MS treatments (non-symptomatic) within specified periods before enrollment;
* an infection requiring systemic anti-infective treatment or vaccination with a live vaccine within 1 month before enrollment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Cumulative number of new gadolinium-enhancing MRI lesions during double-blind treatment period

SECONDARY OUTCOMES:
No. of new active MRI lesions; no. of patients with >=1 objective/subjective MS attack; total no. of MS attacks; no. of patients requiring systemic corticosteroids; change from baseline to wk 12 in EDSS

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Sofia, Bulgaria
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Greenfield Park, Quebec
  - Hull, Quebec
- Czechia (3):
  - Hradec Králové
  - Ostrava
  - Prague
- Germany (4):
  - Marburg
  - Regensburg
  - Tübingen
  - Ulm
- Poland (5):
  - Gdansk
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- Russia (3):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Nitra
- Spain (4):
  - Barcelona
  - Madrid
  - Málaga
  - Seville
- United Kingdom (4):
  - Liverpool
  - Newcastle upon Tyne
  - Nottingham
  - Sheffield